CLINICAL TRIAL: NCT02529566
Title: Human Autograft Mesenchymal Stem Cell Mediated Stabilization of The Degenerative Lumbar Spine
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Foundation for Spinal Research, Education and Humanitarian Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC-2013
Record Dates: First submitted 2015-03-16; First posted 2015-08-20 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Lumbar Degenerative Disc Disease; Lower Back Pain; Chronic Lower Back Pain
Keywords: Lumbar Degenerative Disc Disease; Degenerative Spinal Conditions; Adjacent Segment Disease; Autologous Bone Marrow; Lower Back Pain; Chronic Lower Back Pain; Stem Cells; Lumbar disk; Mesenchymal Stem Cells; Stabilization; CLBP; Autograft; Allograft; Autograft versus Allograft; Facet Joint; Radicular Pain; Adipose; Disc Replacement; Facet Joint Replacement
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigate the potential of tissue grafting that includes human mesenchymal stem cells in the repair and potential stabilization of the degenerative Lumbar disk and facet joint denovo and at the time of surgical reconstruction. Our hypothesis proposes that stabilization will help restore normal structure and function in the degenerative lumbar spine may decrease chronic low back pain associated with the biomechanical demise of the degenerative disk or facet and may improve the natural history of adjacent segment disease found after spinal surgery.

DETAILED DESCRIPTION:
This study is a prospective cohort clinical study, of tissue grafts containing nucleated adult derived autologous or allograft mesenchymal stem cells delivered via intra-discal or intra-facet injections in subjects with chronic low back pain due to either lumbar degenerative disk disease or degenerative facet disease at one to five lumbar levels from L1 to S1 in patients who have been unresponsive to conservative therapy. A second cohort evaluating the development of adjacent segment disease in the lumbar disk and facet joints after nucleated adult mesenchymal stem cells are delivered via intra-discal or intra-facet injections during surgical treatment of adjacent levels for degenerative pathology in the spine. Traditionally, treatment of degenerative spinal conditions has focused on the reconstruction of damaged tissues within the motion segments of the spine. However, biologic treatment of degenerated spinal components should address the etiology of the disease process as opposed to reacting to symptomatology. Strategies to induce a reparative response within the disk and facet joint focus on rebuilding the chondrocyte population and inducing their production of healthy biomechanical extracellular matrix.. Current models to induce a reparative response include; injection of proteins to stimulate proteoglycan production or inhibit the inflammatory response; transfer of genetic material to cells within the dammed structures; engineering of newly formed tissues ex-vivo for implantation; and finally repopulation of the damaged tissues with cells that can repair the injured structures. Subjects who meet strict inclusion/exclusion criteria will be enrolled in the study for injection of allograft or autologous tissue grafting that includes mesenchymal stem cells into their degenerative lumbar spine and followed for a minimum of 2 years for efficacy and adverse events. This is a prospective clinical study cohort comparing allograft to autograft cellular tissue graft injections in subjects with chronic low back pain due to either lumbar degenerative disk disease or degenerative facet disease at one to five lumbar levels from L1 to S1 in patients who have been unresponsive to conservative therapy for at least 3 months.Pre-treatment imaging criteria including Pfirmann Lumbar disk Scores and/or Fujiwara Facet Joint Scores will be noted during the screening visits. After the screening and treatment visits, each subject will be evaluated at 2 weeks, 6 weeks, and again at 3, 6, 12, 24 months after injection.

MRI scanning will be performed at the 6 month post-procedure visit and Pfirmann or Fujiwara Scores will be calculated along with notation of adjacent level disease, epidural pathology (i.e. new disk herniations), or new imaging findings. Patients will be given informed consent to participate the individual treatment they are to receive. This informed consent will follow US FDA guidelines detailed in ICH E6 Section 4.8 of the US Department of Health and Human Services Center for Drug/Biologics Evaluation and Research. At completion of enrollment patients will have surgical sterile preparation and draping. All JCAHO Surgical Care Improvement Project protocols including pre-operative antibiotics will be adhered to. The disk or facet joint of interest will be verified by fluoroscopy and will be sterilely cannulated with an 21 to 11G needle based on anatomic requirements. At this point injection of FDA approved allograft or autograft mesenchymal stem cells within a demineralized bone matrix or hyalouronic acid carrier respectively will be injected in to the facet joint or disk space. Needle will be removed and sterile dressing will be placed. Patients will be placed in a post operative brace for stabilization of the index level to aid in healing. Patients will be discharged home once standard outpatient discharge criteria are met per JCAHO guidelines. Follow up periods will be adhered to as noted above. Patient safety will be strictly monitored in the pre-procedure, peri-procedure, and post-procedure periods for a minimum of 2 years. All patients will be assigned to a follow up surgeon at specific follow up periods and no patients will be denied any care during that period. Physical examination will be documented at each visit. Additionally, scheduled imaging studies will be performed throughout the study period to follow safety. Patients will be followed by their surgical investigator, who will be responsible for diagnosis and management of any complications or adverse events. Development of additional non-spinal disease processes will also be documented to follow any trends that occur including any new related or un-related diseases. Safety of patient confidentiality is an additional study related risk, which will be optimized to the fullest by adhering to the US Health Insurance Portability and Accountability Act of 1996 (HIPAA). Any Serious Adverse Events (SAE) as defined by the US FDA will be reported immediately to the IRB for evaluation. A SAE is classified as an adverse event that results in hospital admission or hospital stay, or alteration of the body in a permanent way. Surgeon investigators will provide pre-operative, peri-operative, and post-operative care for all subjects.

Pre-operative, peri-operative, and post operative data will be collected. Patients will be followed for a minimum of 2 years within the US or Canada with a study investigator for data collection at 2 weeks (±1 wk), 6 weeks (±2 wks), and 3 months (±2 wks), 6 months (±1 mo), 9 months (± 1.5 months), 12 months (±2 mos), and 24 months (±2 mos). Data may be entered as at additional time points as needed. Re-admission, re-injection, and additional hospital/outpatient events will be collected including possible additional surgical procedures. Data will be managed by the investigator or their designee in a computerized database accessible only by research staff with original information kept with the patient medical record in the hospital or follow up sub-investigator office. Comparative statistical analysis will be performed prior to any publication to validate data and conclusions. Study staff and the Principle Investigator (PI) agree to conduct the study(ies) in accordance with the relevant, current protocol(s) and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects. The PI agrees to personally conduct or supervise the described investigation(s). The PI agrees to inform any patients, or any persons used as controls, when drugs or devices are being used for investigational purposes and the PI will ensure that the requirements relating to obtaining informed consent in US 21 CFR Part 50 and institutional review board (IRB) review and approval in US 21 CFR Part 56 are met. The PI agrees to report to the sponsor adverse experiences that occur in the course of the investigation(s) in accordance with US 21 CFR 312.64. The PI understands the potential risks and side effects of all treatments, investigational and standard of care. The PI agrees to ensure that all associates, colleagues, and employees assisting in the conduct of the study(ies) are informed about their obligations in meeting the above commitments. The PI agrees to maintain adequate and accurate records in accordance with US 21 CFR 312.62 and to make those records available for inspection in accordance with US 21 CFR 312.68 if the study is applied and accepted for US FDA review. The PI will ensure that the IRB complies with the requirements of US 21 CFR Part 56 will be responsible for the initial and continuing review and approval of the clinical investigation. The PI also agrees to promptly report to the IRB all changes in the research activity and all unanticipated problems involving risks to human subjects or others. Additionally, the PI will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects. The PI agrees to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements in US 21 CFR Part 312. Medical Ethics are of primary importance during a study of that exposes humans to a new treatment. The scientific merit of the study protocol, potential social value of the research, skill and experience of the investigators, and potential financial exploitation of the study subjects are all of paramount concern. Thus, in addition to abiding by the US FDA Quality Assurance Policy (Form 1572), the World Health Organization's "Declaration of Helsinki" involving the Ethical Principles for Medical Research Involving Human Subjects will be abided by throughout the trial. Finally, as this study involves subjects that reside within the United States, the investigators in this trial will also abide by Title 45 Part 46 of the Code of [US] Federal Regulations, Protection of Human Subjects (45 CFR 46).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, at least 18 years of age, who is unresponsive to conservative therapy and needs surgical reconstruction of the degenerative lumbar spine.

Exclusion Criteria:

* Females who are pregnant or nursing, or plan on becoming pregnant during the 1st year after the procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the age of 18-85 years who presents problems of degenerative lumbar disk.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Screening to 24 months
Oswestry Disability Index (ODI) | Screening to 24 months

SECONDARY OUTCOMES:
SF-12 Health Survey | Screening to 24 months
EQ-5D Quality Adjusted Life Years | Screening to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Farhan N Siddiqi, MD, Principal Investigator — Foundation For Spinal Research Education And Humanitarian Care
Locations (1):
- Trinity Stem Cell Institution, Odessa, Florida, United States